CLINICAL TRIAL: NCT04578327
Title: Investigation of Embodiment for Upper Limb Amputees
Acronym: NISRL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3282-W; 1IK2RX003282-01A2 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-10-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Amputation
Keywords: amputation; sensation; neural interface

STUDY DESIGN:
Intervention Model Description: Aim 1 - An experiment will take place grouped by the type of prosthesis used by upper limb amputees Aim 3 - An experiment will take place grouped by type of sensory restoration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Aim 1 (Experimental): Data from Specific Aim 1 will be used to test the following hypotheses: H1a. The body-powered prosthetic devices are embodied more than passive and myoelectric prosthetic devices. H1b. Passive cosmetic devices are embodied less than actuated cosmetic devices (agency). H1c. Body-powered terminal devices are embodied less than myoelectric terminal devices (agency).
  Interventions: Device: Prosthetic hand
- Aim 3 (Experimental): Data from Specific Aim 3 will be used to test the following hypotheses: H3a. The maximum number of channels elicits more embodiment than the minimum number. H3b. The sensory feedback from passive spatial locations of the hand increases the embodiment compared to sensory feedback just from the grasping spatial locations.
  Interventions: Procedure: Peripheral Nerve Interface

INTERVENTIONS:
Device: Prosthetic hand — Different types of conventional prosthetic limbs will be used by subjects.
  Arms: Aim 1
Procedure: Peripheral Nerve Interface — Different types of peripheral nerve stimulation will take place
  Arms: Aim 3

SUMMARY:
Today, prosthetic hands are numb. They provide no tactile or proprioceptive sensory information back to the user. The lack of sensory feedback has been shown to reduce the utility of a prosthesis by half. The prosthesis is seen as a tool, not as an incorporated part of the body schema. Only now are there chronically-implantable technologies which can provide physiologically appropriate sensory feedback to upper limb amputees to recreate tactile and proprioceptive percepts. These sensations are the building blocks to enable the embodiment of the device. Furthermore, newly developed outcome measures are now available which can detail the improved embodiment such neural interfaces can create. The investigator's mission is to enable the embodiment of artificial devices using peripheral nerve stimulation and thereby close the gap between the experience of our intact physiological systems and those using prosthetic remedies.

This investigation of embodiment for upper limb amputees is organized into three main areas of work including 1) normative data collection, 2) device development, and 3) characterization of embodiment using peripheral nerve stimulation. The normative data collection will quantify the embodiment of conventional cosmetic, body-powered, and myoelectric prosthetic hand options using a modified Rubber Hand Illusion protocol (Specific Aim 1). This thrust will ask how does the amount of embodiment vary among conventional prosthetic hands as well as probe the relationship between agency and embodiment. The device development project entails the design of multi-modal sensors in order to study full-hand embodiment (Specific Aim 2). The ability to measure and then elicit sensation on the passive surfaces of the hand (palm, ulnar border, and dorsal surface) has never been explored. Here, a multi-modal sensor which can detect proximity, contact, and force will be integrated into a commercially available prosthetic hand in order to provide detailed measurements across the palm, ulnar border, and dorsal surfaces in order to study embodiment in more depth. Finally, the characterization of embodiment using peripheral nerve stimulation will take place over a multiple subject factorial experiment which quantifies the effects of quantity and spatial parameters of the peripheral nerve stimulation on the embodiment of prosthetic hands (Specific Aim 3). This study asks what somatosensory percepts from the hand are most critical for embodiment by varying the parameters of the peripheral nerve stimulation (quantity and spatiality) and measuring the level of embodiment in each case.

DETAILED DESCRIPTION:
Leveraging advancements in neural interfaces, biomechatronic devices, and myoelectric control algorithms, my research mission is to enable the embodiment of artificial devices by providing physiologically appropriate somatosensory feedback.

Specific Aim 1: How does the amount of embodiment vary among conventional prosthetic hands?.

Data from Specific Aim 1 will be used to test the following hypotheses: H1a. The body-powered prosthetic devices are embodied more than passive and myoelectric prosthetic devices. H1b. Passive cosmetic devices are embodied less than actuated cosmetic devices (agency). H1c. Body-powered terminal devices are embodied less than myoelectric terminal devices (agency).

Specific Aim 2: Design of Multi-Modal Sensors for Full Hand Sensation (No human subject experiments.) Specific Aim 3: What somatosensory percepts from the hand are most critical for embodiment? Data from Specific Aim 3 will be used to test the following hypotheses: H3a. The maximum number of channels elicits more embodiment than the minimum number. H3b. The sensory feedback from passive spatial locations of the hand increases the embodiment compared to sensory feedback just from the grasping spatial locations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be either able bodied or have an upper limb difference.
* Both Veterans and non-Veterans will be eligible.

Exclusion Criteria:

* No other musculoskeletal injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Southampton Hand Assessment Procedure | Through study completion, an average of 1 year
  Scores the ability of the user to perform activities of daily living using the prosthetic system.
Patient Experience Measure | Through study completion, an average of 1 year
  Assesses the subject's perspective on the embodiment of the prosthetic system. The Patient Experience Measure (PEM) is a validated outcome measure which uses a survey to identify the experience of the person with amputation. The qualitative and quantitative survey produces outcome measures identifying the patient experience across multiple modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob L. Segil, PhD MS, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No